CLINICAL TRIAL: NCT01581645
Title: Increasing Mobility in Parkinsonian Patients With Freezing of Gait and Gait Hypokinesia With an Adjustable, Attachable Laser (Mobilaser)
Brief Title: Mobilaser Study to Help With People Who Are Having Problems With Their Gait
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jay A. Van Gerpen, Assistant Professor of Neurology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-002978
Record Dates: First submitted 2011-11-10; First posted 2012-04-20 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease; Parkinsonism
Keywords: Parkinson's disease; Parkinsonism; Gait problems; Freezing gait
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Mobility Limitation | interventions — Lasers; Walkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobilaser (Experimental): Patients will begin by collecting data at home without using the mobilaser. They will then be given the mobilaser to use at home for 6 weeks while they collect data on whether their gait has improved. They will then have to return the Mobilaser to the clinic and collect data at home for 3 days to see if there is a difference.
  Interventions: Device: Mobilaser

INTERVENTIONS:
Device: Mobilaser — Patients will begin by collecting data at home without using the mobilaser. They will then be given the mobilaser to use at home for 6 weeks while they collect data on whether their gait has improved. They will then have to return the Mobilaser to the clinic and collect data at home for 3 days to see if there is a difference.
  Other Names: Laser; Walker with laser

SUMMARY:
Does use of the Mobilaser reduce freezing of gait (FOG) and stride reduction in patients with Parkinson's disease and Parkinsonism.

DETAILED DESCRIPTION:
Can patients walk faster and have less freezing when using the mobilaser then when not using it

ELIGIBILITY:
Inclusion Criteria:

* Parkinsonian patients with Freezing of Gait or Gait hesitation.
* Must have evidence of bradykinesia ambulating (stride reduction or reduced arm swing)
* Must have a constant caregiver

Exclusion Criteria:

* No cardiopulmonary contraindications to ambulation, e.g., unstable angina pectoris;
* Severe arthritis;
* Cerebellar or sensory ataxia;
* Recent knee or hip surgery

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Gait | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay Van Gerpen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States